CLINICAL TRIAL: NCT06806488
Title: Retrospective Observational Study to Assess Clinical Characteristics and Outcome of Patients with Marginal Zone Lymphomas
Brief Title: Study to Assess Clinical Characteristics and Outcome of Patients with Marginal Zone Lymphomas
Acronym: MarZoLyOss
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: MarZoLyOss
Record Dates: First submitted 2024-12-03; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-10

CONDITIONS: Marginal Zone B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a purely retrospective and observational monocentric study

DETAILED DESCRIPTION:
the study aimed at describing the characteristics and outcome of Marginal zone lymphoma patients who were diagnosed and treated in our Hospital between December 2012 and December 2018

ELIGIBILITY:
Inclusion Criteria:

1. Marginal zone lymphoma patients who were diagnosed and treated in our Hospital between December 2012 and December 2018.
2. Age ≥ 18 years at enrolment.
3. Written informed consent (if applicable)

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Marginal zone lymphoma patients who were diagnosed and treated in our Hospital between December 2012 and December 2018
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
clinical characteristics of Marginal zone lymphoma patients | through study completion, an average of 1 years
  to descrive clinical characteristics of Marginal zone lymphoma patients who were diagnosed and treated in our Hospital.

SECONDARY OUTCOMES:
effectiveness | through study completion, an average of 1 years
  It includes:
  1. Description of treatment duration and causes of treatment discontinuation.
  2. Description of adverse events / safety of the treatments
  3. Assessment of patients' survival.
  4. Description of the medical resource utilization, including number of emergency department visits, hospitalizations, use of hematopoietic growth factors and antibiotics, and blood product transfusions.
  5. Patient clinical and biological characteristics and disease biological profile at baseline of Marginal zone lymphoma cases
safety | through study completion, an average of 1 years
  It includes:
  1. Description of treatment duration and causes of treatment discontinuation.
  2. Description of adverse events / safety of the treatments
  3. Assessment of patients' survival.
  4. Description of the medical resource utilization, including number of emergency department visits, hospitalizations, use of hematopoietic growth factors and antibiotics, and blood product transfusions.
  5. Patient clinical and biological characteristics and disease biological profile at baseline of Marginal zone lymphoma cases

CONTACTS AND LOCATIONS:
Overall Officials: Pier Luigi Zinzani, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero - Universitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No